CLINICAL TRIAL: NCT04756063
Title: Parenteral Ascorbic Acid Repletion in TransplantatIon (PARTI): A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Parenteral Ascorbic Acid Repletion in TransplantatIon
Acronym: PARTI
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Resources
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-1153; A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY (Other: UW Madison); Protocol Version 12/5/2024 (Other: UW Madison)
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Liver Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ascorbic Acid (AA) (Experimental): The first intravenous dosage of 1500mg of AA in 100mL of normal saline (NS) will be administered after induction of general anesthesia and invasive line placement prior to surgical incision. An identical dosage will be delivered approximately every 6 hours for the first 48 hours, for a total of 8 doses
  Interventions: Drug: Ascorbic acid
- Placebo (Placebo Comparator): The first intravenous dosage of placebo (100 mL of NS) will be administered after induction of general anesthesia and invasive line placement prior to surgical incision. An identical dosage will be delivered approximately every 6 hours for the first 48 hours, for a total of 8 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ascorbic acid — Intravenous vitamin C
  Other Names: vitamin C; ASCOR
  Arms: Ascorbic Acid (AA)
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
A single-center, randomized, double-blinded placebo-controlled trial is proposed to investigate administration of supraphysiologic doses of ascorbic acid (vitamin C, AA) to patients undergoing liver transplantation. Participants randomized to the intervention group will receive intravenous (IV) AA 1500 mg every 6 hours for 48 hours. Participants randomized to the control group will receive a saline placebo. The primary study outcome will be a change in the Sequential Organ Failure Assessment (SOFA) score from baseline to three days after the first dose of drug (dSOFA3). Secondary outcomes will include total vasopressor dose in norepinephrine equivalents, 30-day and 1-year mortality, and serum AA levels.

DETAILED DESCRIPTION:
HYPOTHESIS: Administration of supraphysiologic doses of parenteral AA in the perioperative period for patients undergoing liver transplantation will improve Sequential Organ Failure Assessment (SOFA) scores, vasopressor usage and biochemical, cellular and clinical end-organ damage.

Specific Aim: Determine the clinical response to parenteral AA supplementation in patients undergoing liver transplantation by a randomized, double-blinded, placebo-controlled clinical trial.

Study Design: This study is a prospective, single-center, randomized trial in which 90 participants will be enrolled at the University of Wisconsin Hospitals and Clinics (UWHC). Participants must meet study eligibility criteria and be scheduled to undergo primary deceased donor solitary liver transplantation. Participants will be randomized to receive 8 doses of 1500 mg AA IV or volume-equivalent placebo every 6 hours for 48 hours, in addition to standard medical management.

ELIGIBILITY:
Inclusion Criteria:

* The subject is scheduled to undergo primary deceased donor solidary liver transplantation

Exclusion Criteria:

* Non-English speaking
* Known or believed to be pregnant
* Subject is a prisoner
* Impaired decision-making capacity (i.e., current encephalopathy)
* Known allergy to AA
* Concurrent organ transplantation (i.e., simultaneous liver-kidney transplantation)
* Planned veno-venous bypass use in the operating room
* Prior parenteral or oral AA repletion
* History of nephrolithiasis or oxaluria
* Vitamin C supplement use or administration (including HAT therapy) within the last month prior to transplantation
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Sickle cell anemia
* Hereditary hemochromatosis
* Preoperative anuria or creatinine >2.5mg/dL in patient not on renal replacement therapy
* Current enrollment in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Change in Sequential Organ Failure Assessment (SOFA) Score | baseline to 3 days after first dose
  SOFA scores are a widely used composite measure of multiorgan dysfunction, validated as an accurate predictor of short- and long-term mortality in the general ICU and liver transplant populations. Change in SOFA from baseline (delta SOFA or dSOFA) has been shown to be more predictive of mortality than other derivatives such as absolute interval SOFA scores and has been recommended as the preferred endpoint in critical care settings
  The total possible range of scores is 0-24, higher scores are indicative of a higher degree of dysfunction.

SECONDARY OUTCOMES:
Serum AA Levels | Pre-treatment (baseline) and Post-treatment (up to 1 week)
Total Vasopressor Dose in Norepinephrine Equivalents per Kilogram | from start of anesthesia (day 1) to end of ICU stay (up to 1 week)
Incidence of Early Graft Dysfunction | postoperative (up to 7 days or until discharge, whichever came first)
  As defined per Olthoff as: total bilirubin ≥10 or INR≥1.6 on day 7, or transaminase >2000 within first 7 days
Postoperative Day 7 SOFA Score | postoperative (up to 3 days)
  Total range of scores 0-24 where higher scores indicate higher dysfunction.
Days on Ventilator | postoperative (up to ~ 7 days)
Incidence of Infection | postoperative (up to ~ 7 days)
  Surgical site, bloodstream & intra-abdominal infection rates
Length of ICU stay | postoperative (up to ~ 7 days)
Length of Hospital stay | postoperative (up to ~ 30 days)
30 day Mortality | up to 30 days post-op
1-year Mortality | up to 1-year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Molly Groose, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers up to 7 years after the completion of the primary endpoint by contacting Dr. Molly Groose, the Principal Investigator of this study
Supporting Information: Study Protocol
Time Frame: up to 7 years after primary completion